CLINICAL TRIAL: NCT02855944
Title: ARIEL4 (Assessment of Rucaparib In Ovarian CancEr TriaL): A Phase 3 Multicenter, Randomized Study of Rucaparib Versus Chemotherapy in Patients With Relapsed, BRCA Mutant, High Grade Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: ARIEL4: A Study of Rucaparib Versus Chemotherapy BRCA Mutant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-043; 2016-000816-14 (EudraCT Number)
Record Dates: First submitted 2016-07-22; First posted 2016-08-04 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: ovarian cancer; fallopian tube cancer; primary peritoneal cancer; peritoneal cancer; platinum sensitive; relapsed disease; PARP Inhibitor; PARP; rucaparib; ruca; homologous recombination; homologous recombination deficiency; genomic scarring; loss of heterozygosity; CO-338; PF-01367338; PF 01367338; CO-338-043; platinum sensitive ovarian cancer; platinum sensitive fallopian tube cancer; platinum sensitive primary peritoneal cancer; platinum sensitive peritoneal cancer; gynecological cancer; Clovis; Clovis oncology; ARIEL2; ARIEL 2; ARIEL-2; ARIEL-3; ARIEL 3; ARIEL3; ARIEL4; ARIEL-4; ARIEL 4; A4; advanced OC; platinum resistant ovarian cancer; platinum resistant primary ovarian cancer; Rubraca; High grade serous; Partially platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Recurrence | interventions — Drug Therapy; Cisplatin; Carboplatin; CP protocol; Gemcitabine; Paclitaxel; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rucaparib (Experimental): Drug: Oral rucaparib
  600 mg BID (twice a day)
  Other Names:
  * CO-338
  * PF 01367338
  * AG 14699
  * Rubraca
  Interventions: Drug: Rucaparib
- Chemotherapy (Active Comparator): Monotherapy platinum (cisplatin or carboplatin) or platinum-based doublet chemotherapy (carboplatin/paclitaxel, carboplatin/gemcitabine, or cisplatin/gemcitabine administered per local standard of care and regulations. Specific comparator will depend on platinum status and investigator decision.
  Single agent paclitaxel will be administered per local standard of care and regulations. Specific comparator will depend on platinum status and investigator decision.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy will be administered per local standard of care and regulations. Specific comparator will depend on platinum status and investigator decision.
  Other Names: Cisplatin; carboplatin; carboplatin/paclitaxel; carboplatin/gemcitabine; paclitaxel
  Arms: Chemotherapy
Drug: Rucaparib — Tablets of rucaparib, at a dose of 600 mg, will be taken orally twice a day
  Other Names: CO-338; AG 14699; PF 01367338; Rubraca
  Arms: Rucaparib

SUMMARY:
The purpose of this study is to determine how patients with ovarian, fallopian tube, and primary peritoneal cancer will best respond to treatment with rucaparib versus chemotherapy.

DETAILED DESCRIPTION:
Rucaparib is an orally available, small molecule inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) being developed for treatment of ovarian cancer associated with homologous recombination (HR) DNA repair deficiency (HRD). The safety and efficacy of rucaparib has been evaluated in several Phase 1 and Phase 2 studies. An oral formulation is the focus of current development efforts. Rucaparib is currently being investigated as monotherapy in patients with cancer associated with breast cancer susceptibility gene 1 (BRCA1) or BRCA2 mutations.

While PARP inhibitors have demonstrated consistent robust clinical activity in patients with relapsed ovarian cancer associated with HRD, prospective studies evaluating efficacy and safety of PARPi versus standard of care chemotherapy have been limited. The primary purpose of this Phase 3 study is to compare the efficacy and safety of rucaparib versus chemotherapy as treatment for relapsed ovarian cancer in patients with a deleterious BRCA1/2 mutation in their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age at the time the informed consent form is signed
* Have a histologically confirmed diagnosis of high-grade serous or Grade 2 or Grade 3 endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Received ≥ 2 prior chemotherapy regimens and have relapsed or progressive disease as confirmed by radiologic assessment
* Have biopsiable and evaluable disease. Note: biopsy is optional for patients known to harbor a BRCA1/2 mutation
* Have sufficient archival formalin-fixed paraffin-embedded (FFPE) tumor tissue available for planned analyses

Exclusion Criteria:

* History of prior cancers except for those that have been curatively treated, with no evidence of cancer currently (provided all chemotherapy was completed >6 months prior and/or bone marrow transplant >2 years prior to first dose of rucaparib).
* Prior treatment with any PARP inhibitor
* Symptomatic and/or untreated central nervous system metastases
* Pre-existing duodenal stent and/or any other gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of rucaparib
* Women who are pregnant or breast feeding
* Hospitalization for bowel obstruction within 3 months prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (2):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Augusta University, Augusta, Georgia
- Brazil (8):
  - Hospital Haroldo Juacaba Instituto do Cancer do Ceara, Fortaleza, Ceará
  - Instituto de Oncologia do Parana (IOP), Curitiba, Paraná
  - União Brasileira de Educação e Assistência / Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - CEPON-Centro de pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Hospital do Cancer de Barretos, Barretos, São Paulo
  - Instituto Nacional de Câncer Hospital do Câncer II, Rio de Janeiro
  - Hospital Pérola Byington - Centro de Referência da Saúde da Mulher, São Paulo
  - Hospital São Camilo, São Paulo
- Canada (5):
  - Tom Baker Cancer Center, Calgary, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal (CHUM), Montreal, Quebec
  - CIUSSS de l'Estrie CHUS, Sherbrooke, Quebec
- Czechia (4):
  - Masarykuv Onkologicky Ustav, Oddeleni komplexni klinicke onkologie, Brno, Jihormoravsky KRAJ
  - Fakultni Nemocnice v Motole, Prague, Prague
  - Fakultní Nemocnice Ostrava, Ostrava
  - Všeobecná Fakultní Nemocnice v Praze, Prague
- Hungary (2):
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Országos Onkológiai Intézet, Budapest
- Israel (6):
  - Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Oncology Dept., Tel Aviv
- Italy (8):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Istituto per la Ricerca e la Cura del Cancro Istituto di Candiolo, Candiolo
  - AO per l'emergenza Cannizzaro, Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Istituto Nazionale per lo studio e la cura dei tumori "Fondazione Pascale" Oncologia Medica, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Poland (6):
  - Niepubliczny Zaklad Opieki Zdrowotnej Innowacyjna Medycyna Sp z o.o., Grzybnica, West Pomeranian Voivodeship
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie, Bialystok
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Pozna, Poznan
  - Pomorska Akademia Medyczna w Szczecinie, Samodzielny Publiczny Szpital Kliniczny Nr 2, Szczecin
- Russia (12):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Kursk Regional Oncologic Dispensary, Kursk
  - Moscow Clinical Scientific and Practical Center of Moscow Healthcare Department, Moscow
  - Omsk Region Clinical Oncologic Dispensary, Omsk
  - Pyatigorsk Oncological Dispensary, Pyatigorsk
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Pavlov First Saint-Petersburg State Medical University, Saint Petersburg
  - Saint Petersburg City Oncological Dispensary, Saint Petersburg
  - State Healthcare Institution Oncologic Dispensary No. 2 - Health Department of Krasnodar Region, Saint Petersburg
  - Republican oncological dispensary of Republic of Mordovia, Saransk
  - State Healthcare Institution Oncologic Dispensary No. 2 - Health Department of Krasnodar Region, Sochi
  - Republic Clinical Oncology Dispensary of the Ministry of Healthcare of Republic of Bashkortostan, Ufa
- Spain (8):
  - Centro Oncologico Regional de Galicia, A Coruña
  - Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Vall DHebron, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Cancer Center, Madrid
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario La Paz, Madrid
- Ukraine (6):
  - Dnipropetrovsk City Multifield Clinical Hospital Number 4, Dnipropetrovsk
  - National Cancer Institute of the Ministry of Health of Ukraine, Kyiv
  - Volyn Regional Oncology Dispensary, Lutsk
  - Lviv Regional Oncology Dispensary, Lviv
  - Sumy Regional Oncology Center, Sumy
  - Zakarpattya Regional Clinical Oncological Dispensary, Uzhhorod
- United Kingdom (10):
  - The Christie NHS Foundation Trust - Clinical Trial Pharmacy, Manchester, England
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre NHS Trust, Cardiff
  - University Hospital of Coventry and Warwickshire NHS Trust, Coventry
  - Derby Teaching Hospital NHS Foundation Trust, Derby
  - NHS Greater Glasgow and Clyde, Glasgow
  - University College London Hospitals, London
  - East and North Hertfordshire NHS Trust, Middlesex
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Derived] Oza AM, Lisyanskaya A, Fedenko A, de Melo AC, Shparyk Y, Rakhmatullina I, Bondarenko I, Colombo N, Svintsitskiy V, Biela L, Nechaeva M, Lorusso D, Scambia G, Cibula D, Poka R, Oaknin A, Safra T, Mackowiak-Matejczyk B, Ma L, Thomas D, Lin KK, McLachlan K, Goble S, Kristeleit R. Rucaparib versus chemotherapy for treatment of relapsed ovarian cancer with deleterious BRCA1 or BRCA2 mutation (ARIEL4): final results of an international, open-label, randomised, phase 3 trial. Lancet Oncol. 2025 Feb;26(2):249-264. doi: 10.1016/S1470-2045(24)00674-0. PMID 39914419
- [Derived] Kristeleit R, Lisyanskaya A, Fedenko A, Dvorkin M, de Melo AC, Shparyk Y, Rakhmatullina I, Bondarenko I, Colombo N, Svintsitskiy V, Biela L, Nechaeva M, Lorusso D, Scambia G, Cibula D, Poka R, Oaknin A, Safra T, Mackowiak-Matejczyk B, Ma L, Thomas D, Lin KK, McLachlan K, Goble S, Oza AM. Rucaparib versus standard-of-care chemotherapy in patients with relapsed ovarian cancer and a deleterious BRCA1 or BRCA2 mutation (ARIEL4): an international, open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Apr;23(4):465-478. doi: 10.1016/S1470-2045(22)00122-X. Epub 2022 Mar 14. PMID 35298906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 349 patients from 64 sites across 12 countries were enrolled in the initial Treatment Part of the study and randomized to receive rucaparib or chemotherapy. Patients randomized to chemotherapy had the option to cross over to receive rucaparib in the Crossover Part of the study upon progression of disease.
Groups:
- Rucaparib: Patients randomized to the rucaparib arm received oral rucaparib 600 mg twice a day (BID) in continuous 28-day cycles.
- Chemotherapy: Patients randomized to the chemotherapy arm received either weekly intravenous (IV) paclitaxel or IV platinum-based chemotherapy per investigator choice and per standard of care. The starting dose of weekly paclitaxel was 60 to 80 mg/m2 administered via IV infusion (ie, on Days 1, 8, and 15) in each 28-day cycle (with a week break from dosing on Day 22 in each cycle). The dosage and administration of single-agent cisplatin or carboplatin or doublet carboplatin/paclitaxel, carboplatin/gemcitabine, or cisplatin/gemcitabine IV infusion followed institutional guidelines for each agent. Upon progression of disease, patients had the option to cross over to rucaparib and receive oral rucaparib 600 mg BID in continuous 28-day cycles.
Period: Period 1: Treatment
Arm/Group | Rucaparib | Chemotherapy
Started | 233 | 116
Completed | 218 | 113
Not Completed | 15 | 3
Not completed — Ongoing | 14 | 0
Not completed — Discontinued prior to starting study drug | 1 | 3
Period: Period 2: Crossover to Rucaparib
Arm/Group | Rucaparib | Chemotherapy
Started | 0 | 80
Completed | 0 | 75
Not Completed | 0 | 5
Not completed — Ongoing | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Rucaparib: Patients randomized to the rucaparib arm.
- Chemotherapy: Patients randomized to the chemotherapy arm.
- Total: Total of all reporting groups
Arm/Group | Rucaparib | Chemotherapy | Total
Number analyzed (Participants) | 233 | 116 | 349
Age, Continuous [Median (Full Range); unit: years] | 58.0 [38 to 81] | 58.5 [38 to 85] | 58.0 [38 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 116 | 349
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 219 | 113 | 332
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 1 | 6
ECOG at Baseline [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Scale. ECOG 0 = Fully active, able to carry on all pre-disease performance without restriction. ECOG 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (eg, light house work or office work).
  Participants
    ECOG 0 | 125 | 72 | 197
    ECOG 1 | 108 | 44 | 152
Number of Prior Chemotherapy Regimens [Count of Participants; unit: Participants]
  2 | 134 | 68 | 202
  3 | 58 | 28 | 86
  4 | 23 | 11 | 34
  5 | 7 | 5 | 12
  >5 | 11 | 4 | 15
Number of Prior Platinum Regimens [Count of Participants; unit: Participants]
  1 | 12 | 6 | 18
  2 | 156 | 74 | 230
  3 | 48 | 28 | 76
  4 | 11 | 7 | 18
  5 | 2 | 1 | 3
  >5 | 4 | 0 | 4
Randomization Stratification: Platinum Status [Count of Participants; unit: Participants] — * Platinum resistant: patients who progressed ≥ 1 to < 6 months after the last dose of platinum-based chemotherapy;
  * Partially platinum-sensitive: patients who progressed ≥ 6 to < 12 months after last dose of platinum-based chemotherapy; and
  * Platinum sensitive: patients who progressed ≥ 12 months after last dose of platinum-based chemotherapy
  Participants
    Platinum resistant | 120 | 59 | 179
    Partially platinum-sensitive | 65 | 31 | 96
    Platinum sensitive | 48 | 26 | 74
Combined Local and Central Lab BRCA Mutation Results [Count of Participants; unit: Participants] — * BRCA1: patients with a deleterious breast cancer susceptibility gene 1 (BRCA1) mutation in their tumor
  * BRCA2: patients with a deleterious breast cancer susceptibility gene 2 (BRCA2) mutation in their tumor
  * Non-BRCA: patients without a BRCA mutation in their tumor
  Participants
    BRCA1 | 181 | 79 | 260
    BRCA2 | 52 | 36 | 88
    Non-BRCA | 0 | 1 | 1
Mutation Type [Count of Participants; unit: Participants]
  Germline | 198 | 95 | 293
  Somatic | 35 | 19 | 54
  Not Available | 0 | 2 | 2
Patients with a BRCA Reversion Mutation [Count of Participants; unit: Participants] | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Investigator Assessed Progression-Free Survival (invPFS) by RECIST Version 1.1 for Rucaparib Versus Chemotherapy (Efficacy Population)
Description: The primary efficacy endpoint is invPFS for the Treatment Part of the study. The time to invPFS is calculated in months as the time from randomization to disease progression +1 day, as determined by RECIST v1.1 (Response Evaluation Criteria in Solid Tumors) criteria or death due to any cause, whichever occurs first. Progression is defined using RECIST v1.1, as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessments every 8 weeks from Cycle 1 Day 1 (C1D1) until disease progression, death, or initiation of subsequent treatment. After 18 months on study, assessments every 16 weeks. Total follow-up was up to approximately 3.5 years.
Population: Efficacy Population - All randomized patients in the treatment part of study with a deleterious BRCA mutation, excluding those identified to have a BRCA reversion mutation. As noted in the Baseline Characteristics Module, 1 patient in the Chemotherapy Arm did not have a BRCA mutation (Non-BRCA) and is therefore excluded from the overall number of patients analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 220 | 105
Months | 7.4 [7.3 to 9.1] | 5.7 [5.5 to 7.3]
Statistical Analysis 1: Comparison: Rucaparib vs Chemotherapy; Test type: Superiority; p = 0.0010, Regression, Cox; Cox Proportional Hazard = 0.639, 95% CI 2-sided [0.489 to 0.835]

2. Primary Outcome: Investigator Assessed Progression-Free Survival (invPFS) by RECIST Version 1.1 for Rucaparib Versus Chemotherapy (ITT Population)
Description: as for outcome 1
Time Frame: Assessments every 8 weeks from C1D1 until disease progression, death, or initiation of subsequent treatment. After 18 months on study, assessments every 16 weeks. Total follow-up was up to approximately 3.5 years.
Population: Intent-to-treat (ITT) Population - All randomized patients in the treatment part of study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 233 | 116
Months | 7.4 [6.7 to 7.9] | 5.7 [5.5 to 6.7]
Statistical Analysis 1: Comparison: Rucaparib vs Chemotherapy; Test type: Superiority; p = 0.0017, Regression, Cox; Cox Proportional Hazard = 0.665, 95% CI 2-sided [0.516 to 0.858]

3. Secondary Outcome: Investigator Assessed Overall Response Rate (ORR) by RECIST v1.1 (Efficacy Population)
Description: A secondary endpoint is the ORR for the Treatment Part of the study. ORR is defined as the percentage of patients with a confirmed CR (complete response) or PR (partial response) by RECIST v1.1. The confirmed response is defined as a CR or PR on subsequent tumor assessment at least 28 days after first response documentation. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: as for outcome 2
Population: Efficacy population with measurable disease at baseline. Efficacy population defined as all randomized patients with a deleterious BRCA mutation, excluding those identified to have a BRCA reversion mutation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 211 | 96
percentage of participants | 40.3 [33.6 to 47.2] | 32.3 [23.1 to 42.6]

4. Secondary Outcome: Investigator Assessed Overall Response Rate (ORR) by RECIST v1.1 (ITT Population)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Intent-to-treat (ITT) population with measurable disease at baseline. ITT population defined as all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 224 | 106
percentage of participants | 37.9 [31.6 to 44.7] | 30.2 [21.7 to 39.9]

5. Secondary Outcome: Investigator Assessed Duration of Response (DOR) by RECIST v1.1 (Efficacy Population)
Description: A secondary endpoint is the DOR for the Treatment Part of the study. The DOR as assessed by investigator is analyzed in the subgroup of patients who had a confirmed response by RECIST v1.1. DOR for any confirmed RECIST CR or PR will be measured from the date of the first response until the first date that progressive disease (PD) is documented. DOR is calculated in months as the time from the first date of the scan showing a response to the first scan with disease progression +1 day. Any patients with an ongoing response are censored at the date of the last post-baseline scan. Only tumor scans up to and within 6 weeks of start of any subsequent anti-cancer treatment are included. Progressive disease (PD) is defined using RECIST v1.1, as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 2
Population: Efficacy population with measurable disease at baseline and a confirmed response. Efficacy population defined as all randomized patients with a deleterious BRCA mutation, excluding those identified to have a BRCA reversion mutation. As noted in the Baseline Characteristics Module, 1 patient in the Chemotherapy Arm did not have a BRCA mutation (Non-BRCA) and is therefore excluded from the overall number of patients analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 85 | 31
months | 9.4 [7.5 to 11.1] | 7.2 [4.0 to 11.4]
Statistical Analysis 1: Comparison: Rucaparib vs Chemotherapy; Test type: Superiority; p = 0.0401, Regression, Cox; Cox Proportional Hazard = 0.589, 95% CI 2-sided [0.356 to 0.976]

6. Secondary Outcome: Investigator Assessed Duration of Response (DOR) by RECIST v1.1 (ITT Population)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Intent-to-treat (ITT) population with measurable disease at baseline and a confirmed response. ITT population defined as all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 85 | 32
months | 9.4 [7.5 to 11.1] | 7.2 [3.9 to 9.4]
Statistical Analysis 1: Comparison: Rucaparib vs Chemotherapy; Test type: Superiority; p = 0.0240, Regression, Cox; Cox Proportional Hazard = 0.564, 95% CI 2-sided [0.343 to 0.927]

7. Secondary Outcome: Investigator Assessed Overall Response Rate (ORR) by RECIST v1.1 and/or CA-125 Response (Efficacy Population)
Description: A secondary endpoint is ORR for the Treatment Part of the study defined as the percentage of patients with best response of CR or PR using RECIST v1.1 or response per Gynecologic Cancer InterGroup Cancer Antigen 125 (GCIG CA-125) criteria. Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Response to CA-125 has occurred if there is at least a 50% decrease from baseline: 1. in a sample collected after initiation of study treatment AND 2. that is confirmed in a subsequent sample collected ≥21 days after the prior sample. The absolute value of this confirmatory sample must be ≤110% of the prior sample. The date when the first sample with a 50% decrease from baseline is observed is the date of the CA-125 response.
Time Frame: as for outcome 2
Population: Efficacy population with measurable disease at baseline and/or CA-125 response evaluable. Efficacy population defined as all randomized patients with a deleterious BRCA mutation, excluding those identified to have a BRCA reversion mutation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 217 | 101
percentage of patients | 50.7 [43.8 to 57.5] | 43.6 [33.7 to 53.8]

8. Secondary Outcome: Investigator Assessed Overall Response Rate (ORR) by RECIST v1.1 and/or CA-125 Response (ITT Population)
Description: as for outcome 7
Time Frame: as for outcome 2
Population: Intent-to-treat (ITT) population with measurable disease at baseline and/or CA-125 response evaluable. ITT population defined as all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 230 | 111
percentage of patients | 47.8 [41.2 to 54.5] | 40.5 [31.3 to 50.3]

9. Secondary Outcome: Least Squares Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status Score for the First 6 Cycles (Efficacy Population)
Description: EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer patients. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. Mean changes from baseline global score over the first 6 cycles in the Treatment Part of the study were analyzed.
Time Frame: Baseline to the end of Cycle 6, or up to approximately 6 months
Population: Efficacy population - All randomized patients with a deleterious BRCA mutation, excluding those identified to have a BRCA reversion mutation, and with a baseline value and at least one post-baseline value for the EORTC QLQ-C30 Global Health Status score during the first 6 cycles.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 197 | 91
score on a scale | 0.5 (0.55) | 0.3 (0.86)

10. Secondary Outcome: Least Squares Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status Score for the First 6 Cycles (ITT Population)
Description: as for outcome 9
Time Frame: Baseline to the end of Cycle 6, or up to approximately 6 months
Population: Intent-to-treat (ITT) population - All randomized patients with a baseline value and at least one post-baseline value for the EORTC QLQ-C30 Global Health Status score during the first 6 cycles.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 207 | 101
score on a scale | 0.6 (0.54) | 0.4 (0.82)

11. Secondary Outcome: Overall Survival (Efficacy Population)
Description: Overall survival (OS) is defined as the number of days from the date of randomization to the date of death (due to any cause). Patients who are still alive were censored on the date of their last available visit or last date known to be alive.
Time Frame: All patients were followed for survival up to approximately 3.5 years.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 220 | 105
Months | 21.1 [17.9 to 24.9] | 26.2 [22.2 to 29.1]

12. Secondary Outcome: Overall Survival (ITT Population)
Description: as for outcome 11
Time Frame: All patients were followed for survival up to approximately 3.5 years.
Population: Intent-to-Treat (ITT) Population - All randomized patients in the treatment part of the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib | Chemotherapy
Number analyzed (Participants) | 233 | 116
Months | 19.4 [15.2 to 23.6] | 25.4 [21.4 to 27.6]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from date of first dose of study drug until 28 days after last dose of study drug, approximately 3.5 years.
Description: Adverse events are reported for the Safety Population, defined as patients who received at least one dose of protocol-specified treatment.
Groups:
- Rucaparib (Treatment Part): Patients randomized to the rucaparib arm in the Treatment Part of the study.
- Chemotherapy (Treatment Part): Patients randomized to the chemotherapy arm in the Treatment Part of the study.
- Rucaparib (Crossover Part): Patients randomized to chemotherapy who then crossed over upon disease progression and were treated with rucaparib.
Arm/Group | Rucaparib (Treatment Part) | Chemotherapy (Treatment Part) | Rucaparib (Crossover Part)
All-Cause Mortality (participants affected / at risk) | 16/232 | 4/113 | 3/80
Serious Adverse Events (participants affected / at risk) | 66/232 | 14/113 | 24/80
Other Adverse Events (participants affected / at risk) | 229/232 | 109/113 | 76/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib (Treatment Part) (N=232) | Chemotherapy (Treatment Part) (N=113) | Rucaparib (Crossover Part) (N=80)
Anemia (Blood and lymphatic system disorders) | 18 | 2 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dolichocolon acquired (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 6 | 0 | 4
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Small intestine obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0
Death (General disorders) | 2 | 0 | 0
General physical health deterioration (General disorders) | 2 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2
Septic shock (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 1
Blood disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0
Meningoencephalitis herpatic (Infections and infestations) | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib (Treatment Part) (N=232) | Chemotherapy (Treatment Part) (N=113) | Rucaparib (Crossover Part) (N=80)
Anaemia (Blood and lymphatic system disorders) | 130 | 36 | 37
Leukopenia (Blood and lymphatic system disorders) | 24 | 20 | 13
Neutropenia (Blood and lymphatic system disorders) | 49 | 30 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 49 | 16 | 14
Sinus tachycardia (Cardiac disorders) | 7 | 6 | 3
Abdominal distension (Gastrointestinal disorders) | 16 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 57 | 20 | 17
Abdominal pain upper (Gastrointestinal disorders) | 22 | 5 | 8
Ascites (Gastrointestinal disorders) | 14 | 2 | 2
Constipation (Gastrointestinal disorders) | 39 | 19 | 15
Diarrhoea (Gastrointestinal disorders) | 51 | 24 | 14
Dyspepsia (Gastrointestinal disorders) | 19 | 7 | 2
Intestinal obstruction (Gastrointestinal disorders) | 12 | 0 | 5
Nausea (Gastrointestinal disorders) | 128 | 38 | 35
Stomatitis (Gastrointestinal disorders) | 11 | 7 | 3
Vomiting (Gastrointestinal disorders) | 82 | 21 | 17
Asthenia (General disorders) | 68 | 27 | 13
Fatigue (General disorders) | 60 | 30 | 17
Oedema peripheral (General disorders) | 13 | 9 | 2
Pyrexia (General disorders) | 25 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 3 | 5
Urinary tract infection (Infections and infestations) | 21 | 5 | 5
Alanine aminotransferase increased (Investigations) | 79 | 12 | 36
Aspartate aminotransferase increased (Investigations) | 75 | 8 | 30
Blood alkaline phosphatase increased (Investigations) | 19 | 3 | 10
Blood bilirubin increased (Investigations) | 22 | 0 | 8
Blood cholesterol increased (Investigations) | 10 | 7 | 8
Blood creatinine increased (Investigations) | 40 | 10 | 18
Blood urea increased (Investigations) | 11 | 5 | 8
Electrocardiogram QT prolonged (Investigations) | 6 | 6 | 6
Electrocardiogram repolarisation abnormality (Investigations) | 3 | 5 | 4
Neutrophil count decreased (Investigations) | 5 | 7 | 2
Weight decreased (Investigations) | 30 | 4 | 7
Decreased appetite (Metabolism and nutrition disorders) | 48 | 20 | 22
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 5 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 15 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 7 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 8 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 4 | 4
Dizziness (Nervous system disorders) | 13 | 9 | 4
Dysgeusia (Nervous system disorders) | 39 | 8 | 11
Headache (Nervous system disorders) | 18 | 6 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 17 | 2
Neurotoxicity (Nervous system disorders) | 1 | 8 | 2
Paraesthesia (Nervous system disorders) | 5 | 10 | 1
Insomnia (Psychiatric disorders) | 21 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 9 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 40 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 10 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 3 | 8
Rash (Skin and subcutaneous tissue disorders) | 13 | 4 | 4
Hypertension (Vascular disorders) | 8 | 7 | 5
Lymphopenia (Blood and lymphatic system disorders) | 10 | 7 | 5
Abdominal pain lower (Gastrointestinal disorders) | 13 | 2 | 4
Erythema (Skin and subcutaneous tissue disorders) | 4 | 2 | 7
Sinus bradycardia (Cardiac disorders) | 3 | 4 | 4
Mucosal inflammation (General disorders) | 7 | 1 | 4
Hypertransaminasaemia (Hepatobiliary disorders) | 9 | 0 | 4
Blood triglycerides increased (Investigations) | 6 | 5 | 4
Creatinine renal clearance decreased (Investigations) | 11 | 3 | 5
Gamma-glutamyltransferase increased (Investigations) | 8 | 0 | 5
Platelet count decreased (Investigations) | 11 | 1 | 4
Weight increased (Investigations) | 0 | 5 | 4
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02855944/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02855944/SAP_001.pdf